CLINICAL TRIAL: NCT05562596
Title: Liquor Oxysterols Concentrations as Biomarkers in Idiopathic Normal Pressure Hydrocephalus
Brief Title: Normal Pressure Hydrocephalus Biomarkers Investigation
Acronym: NORPHY
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Collaborators: AUSL Latina (Unknown)
Responsible Party: Principal Investigator, Luigi Iuliano, Professor of Internal Medicine, University of Roma La Sapienza
Other Study IDs: Hydro2022
Record Dates: First submitted 2022-06-21; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Normal Pressure Hydrocephalus; Cognitive Impairment
Keywords: normal pressure hydrocephalus; neurodegeneration; cognitive impairment; oxysterols; mass spectrometry
MeSH Terms: conditions — Hydrocephalus, Normal Pressure; Cognitive Dysfunction; Nerve Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Liquor (1 mL) specimens are collected before (BF) and at the time of surgery (SG). Samples are snap frozen at -80 °C until analysis. In particular, sample BF is collected at the time of instrumental evaluation for diagnosis by liquor tap, and SG sample taken during surgery, which is made within one month of sample collection BF.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Measurement of oxysterol profile, including 20 molecules, in liquor before and after surgery — Samples are quantitated by deuterium-labeled mass-spectrometry amalysis.

SUMMARY:
Normal Pressure Hydrocephalus (NPH) is a clinical condition that induces cognitive deterioration that can be reverted, at least in part, by introducing ventricular-peritoneal diversion controlled by a miniaturized valve system.

Mechanisms involved in such an improvement of cognitive function after liquor diversion are unknown.

Oxysterols are a family of cholesterol-related compounds having diverse biological functions. Among others, they are involved in cholesterol homeostasis in the brain and are detectable in liquor, potentially impacting neurodegeneration.

NPH is an ideal clinical model to study oxysterol distribution in liquor before and after ventricular-peritoneal diversion.

DETAILED DESCRIPTION:
Normal-pressure hydrocephalus (NPH) is a progressive, chronic, and extremely complex syndrome, firstly described in 1957, which represents the most common form of reversible dementia in the elderly.

The onset of NPH is on average in the seventh decade of life, with a slightly higher prevalence in males, and the Adam-Hakim triad, which includes dementia, urinary incontinence, and gait deviations, constitutes its clinical mainstay.

Clinical manifestations of NPH are hard to notice, especially at the onset, and the patient itself may not grasp the presence of early signs of NPH until a major event - a fall, for example, occurs.

Diagnosis of NPH is made upon clinical and radiological data and on the effectiveness of cerebrospinal fluid (CSF) shunting by ventricular diversion.

Mechanisms involved in the development of NPH are mainly unknown. Oxysterols are sterol compounds congeners of cholesterol with diverse biological properties. Some of them are linked to cholesterol trafficking in the brain - e.g. 24S-hydroxycholesterol (24S-HC) that allows the transport of cholesterol from the brain to the liver, and are supposedly implicated in neurodegenerative diseases. Evaluation of CSF oxysterols concentration in patients diagnosed with NPH constitutes the primary objective of this study.

CSF levels of oxysterols will be evaluated at two key time points: during the diagnostic work-up, via a spinal tap, and during the surgical treatment of NPH, via ventricular diversion.

In particular, within one month of recruitment, patients are evaluated clinically -including brain MR, cognitive function by MMSE, urinary incontinence, and gait deviation, and are subjected to the spinal tap test to meet the criteria of NPH.

Patients eligible for surgery are then subjected, within one month of diagnosis, to ventricular-peritoneal diversion controlled by a miniaturized valve system. This procedure is known to induce impressive amelioration of symptoms, including cognitive ones.

Oxysterol levels are correlated with the degree of cognitive function, i.e. MMSE score before and after surgery. A second sample of oxysterols is collected at the time of surgery from ventricular drainage to look at any potential difference between regional brain oxysterolome, I.,e. peripheral (spinal and central) nervous system.

Oxysterols are quantitatively measured by isotope dilution gas chromatography mass spectrometry. The first objective is to compare oxysterol levels between two different areas of the circulating liquor, i.e. peripheral (spinal site) and central (ventricular site). In this context, the time frame of the two sample collection is set to two months, i.e. surgery is carried out within one month of the diagnostic spinal tap. The second objective is to assess the correlation between oxysterol levels and minimental status examination score.

This study is designed to cast a light on the pathogenesis of NPH and to evaluate the possible correlation between CSF oxysterols concentration and clinical symptoms severity, with a focus on dementia, assessed via cognitive screening tests such as Mini-Mental State Evaluation (MMSE).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of NPH

Exclusion Criteria:

* Patients with a non-performing ASA score to the intervention

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of NPH based on clinical and a diagnostic tap-test
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-10-30 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Oxysterol levels in peripheral and central brain liquor | 2 months
  Comparison between values of quantitative analysis of oxysterols in liquor collected at time of spinal and central liquor obtained at spinal tap and ventricular drainage
Correlation between oxysterol levels in the peripheral and central liquor and MMSE score | 2 months
  Evaluation of potential correlation between oxysterol levels and mini-mental status examination score.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Iuliano, M.D., Principal Investigator — University of Roma La Sapienza; Gianpaolo Petrella, M.D., Principal Investigator — AUSL Latina
Locations (1):
- Goretti Hospital, Latina, LT, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hakim S, Adams RD. The special clinical problem of symptomatic hydrocephalus with normal cerebrospinal fluid pressure. Observations on cerebrospinal fluid hydrodynamics. J Neurol Sci. 1965 Jul-Aug;2(4):307-27. doi: 10.1016/0022-510x(65)90016-x. No abstract available. PMID 5889177
- [Background] Adams RD, Fisher CM, Hakim S, Ojemann RG, Sweet WH. SYMPTOMATIC OCCULT HYDROCEPHALUS WITH "NORMAL" CEREBROSPINAL-FLUID PRESSURE. A TREATABLE SYNDROME. N Engl J Med. 1965 Jul 15;273:117-26. doi: 10.1056/NEJM196507152730301. No abstract available. PMID 14303656
- [Background] Williams MA, Relkin NR. Diagnosis and management of idiopathic normal-pressure hydrocephalus. Neurol Clin Pract. 2013 Oct;3(5):375-385. doi: 10.1212/CPJ.0b013e3182a78f6b. PMID 24175154
- [Background] Hashimoto M, Ishikawa M, Mori E, Kuwana N; Study of INPH on neurological improvement (SINPHONI). Diagnosis of idiopathic normal pressure hydrocephalus is supported by MRI-based scheme: a prospective cohort study. Cerebrospinal Fluid Res. 2010 Oct 31;7:18. doi: 10.1186/1743-8454-7-18. PMID 21040519
- [Background] Mori E, Ishikawa M, Kato T, Kazui H, Miyake H, Miyajima M, Nakajima M, Hashimoto M, Kuriyama N, Tokuda T, Ishii K, Kaijima M, Hirata Y, Saito M, Arai H; Japanese Society of Normal Pressure Hydrocephalus. Guidelines for management of idiopathic normal pressure hydrocephalus: second edition. Neurol Med Chir (Tokyo). 2012;52(11):775-809. doi: 10.2176/nmc.52.775. PMID 23183074
- [Background] Forner Giner J, Sanz-Requena R, Florez N, Alberich-Bayarri A, Garcia-Marti G, Ponz A, Marti-Bonmati L. Quantitative phase-contrast MRI study of cerebrospinal fluid flow: a method for identifying patients with normal-pressure hydrocephalus. Neurologia. 2014 Mar;29(2):68-75. doi: 10.1016/j.nrl.2013.02.016. Epub 2013 May 3. English, Spanish. PMID 23643684
- [Background] Iuliano L, Crick PJ, Zerbinati C, Tritapepe L, Abdel-Khalik J, Poirot M, Wang Y, Griffiths WJ. Cholesterol metabolites exported from human brain. Steroids. 2015 Jul;99(Pt B):189-93. doi: 10.1016/j.steroids.2015.01.026. Epub 2015 Feb 7. PMID 25668615
- [Background] Crick PJ, William Bentley T, Abdel-Khalik J, Matthews I, Clayton PT, Morris AA, Bigger BW, Zerbinati C, Tritapepe L, Iuliano L, Wang Y, Griffiths WJ. Quantitative charge-tags for sterol and oxysterol analysis. Clin Chem. 2015 Feb;61(2):400-11. doi: 10.1373/clinchem.2014.231332. Epub 2014 Dec 15. PMID 25512642
- [Background] Testa G, Staurenghi E, Zerbinati C, Gargiulo S, Iuliano L, Giaccone G, Fanto F, Poli G, Leonarduzzi G, Gamba P. Changes in brain oxysterols at different stages of Alzheimer's disease: Their involvement in neuroinflammation. Redox Biol. 2016 Dec;10:24-33. doi: 10.1016/j.redox.2016.09.001. Epub 2016 Sep 16. PMID 27687218